CLINICAL TRIAL: NCT04574986
Title: Early Prenatal Interview : Throwback to the Hospital of Montpellier's Experience and Description of the Psychiatric Care Pathway of Pregnant Women.
Brief Title: Description of the Psychiatric Care Pathway of Pregnant Women After the Early Prenatal Interview
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0452
Record Dates: First submitted 2020-09-11; First posted 2020-10-05 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Psychiatric Disorder
Keywords: Orientation to a psychiatric follow-up after EPP; Early Prenatal Interview; Psychiatric disorder during pregnancy
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pregnancy and postpartum are recognized as periods of psychic fragility. However, the psychiatric disorders of women that can emerge during these periods are underdiagnosed and have consequences in particular on the development of the child, his relationship with his parents.

The need for an early diagnosis to allow appropriate treatment seems to be essential.

The pregnancy monitoring is centered on the somatic and little on psychological evaluation of the mother and the father.

In this context, the Early Prenatal Interview (EPP) was created through the perinatal plan of 2005-2007 in order to allow a more precise research of the factors of vulnerabilities likely to be predictive of a somatic, psychological or social disorder.

However, until now, only few pregnant women benefited of this interview. In May 2020, EPP became mandatory for all pregnant women. It now seems important to clearly identify the place, function, organization and usefulness of this interview in order to maximize its benefit in the monitoring of pregnancy

DETAILED DESCRIPTION:
First, the investigators will describe the care pathway for pregnant women who have benefited of an early prenatal interview (EPP) between March 2019 and March 2020, namely continued classic follow-up or referral to a child psychiatrist / psychiatrist.

Then, the investigators will define two subgroups within the women oriented towards psychiatric follow-up: those who had this follow-up and those who did not.

Then, the investigators will identify the factors of failure of this referral to psychiatric follow-up and describe the eventual difficulties encountered by the lack of this follow-up.

Finally, the investigators will try to study these observations made with the perspective of maximizing the benefit of the Early Prenatal Interview in the monitoring of pregnancy.

ELIGIBILITY:
Inclusion criteria:

* No opposition from women to participate in the study
* Women over 18
* Women who had an EPP at Montpellier University Hospital between March 2019 and March 2020

Exclusion criteria:

- age < 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women who had an EPP at Montpellier's hospital between March 2019 and March 2020.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Percentage of pregnant women who have been oriented to a psychiatric follow-up after EPP. | 1 day
  Percentage of pregnant women who have been oriented to a psychiatric follow-up after EPP.

SECONDARY OUTCOMES:
Description of the psychiatric care path after Early Prenatal Interview | 1 day
  Description of the psychiatric care path after Early Prenatal Interview so :
  * percentage of pregnant women who were referred to a midwife
  * percentage of pregnant women who were referred to a child psychiatrist
  * percentage of pregnant women who were referred to an adult psychiatrist
  * percentage of pregnant women who were referred to an other follow-up
Identification of potential factors of failure. | 1 day
  Identification of potential factors of failure : In the number of women who were referral to a child psychiatrist / psychiatrist, search the number of women who didn't see the child or adult psychiatrist and try to identify why for each of these women
Number of Participants with difficulties caused by the lack of follow-up | 1 day
  Number of Participants with difficulties caused by the lack of follow-up as :
  Search for each women who were referral to a child or adult psychiatrist ;
  * mode of delivery and term
  * complications of delivery for the baby or mother
  * hospitalization in psychiatry
  * prolongation of stay in the maternity Then compare for these criterias in women who see the child or adult psychiatrist or women who didn't see him and see if the difficulties are more present in women who didn't have the follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Pauline AVIT, resident, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC